CLINICAL TRIAL: NCT00956137
Title: A Randomised Controlled Trial of Ultrasound-assisted Spinal Anaesthesia in Patients With Difficult Anatomical Landmarks.
Brief Title: Ultrasound-assisted Spinal Anaesthesia in Patients With Difficult Anatomical Landmarks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-0190-AE
Record Dates: First submitted 2009-07-17; First posted 2009-08-11 (Estimated); Last update posted 2017-12-04 (Actual); Status verified 2010-01

CONDITIONS: Spinal Anesthesia
Keywords: spinal anesthesia; ultrasound; palpation; knee; hip; surgery; intervertebral space

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound (Experimental): Use of ultrasound to identify vertebral interspaces for needle insertion.
  Interventions: Procedure: Ultrasound guidance
- Palpation (Active Comparator): Use of manual palpation to identify vertebral landmarks and vertebral interspaces for needle insertion.
  Interventions: Procedure: Manual palpation

INTERVENTIONS:
Procedure: Ultrasound guidance — ultrasound imaging
  Arms: Ultrasound
Procedure: Manual palpation — Manual Palpation of vertebra
  Arms: Palpation

SUMMARY:
Spinal anesthesia is the technique of choice in patients undergoing total joint arthroplasty at Toronto Western Hospital (UHN). The most significant predictor of the ease of performance of spinal anesthesia is the quality of palpable surface landmarks (the spinous processes of the lumbar vertebrae). These surface landmarks may be absent, indistinct or distorted in many of the patients presenting for total joint arthroplasty. This is because of obesity, previous spinal surgery, scoliosis and degenerative changes of aging. The investigators have shown in a previous study that a pre-procedural ultrasound scan of the spine can reliably identify an appropriate site for needle insertion in spinal anesthesia, and that this results in a high success rate on the first needle insertion attempt (84% vs 61-64% in published studies). The investigators therefore believe that this ultrasound-assisted technique of spinal anesthesia is extremely useful, especially in patients with poor-quality surface landmarks. However there are no published randomized controlled trials to date that compare the efficacy of the ultrasound-assisted technique with the traditional surface landmark-guided technique of spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Planned spinal anesthesia for elective lower limb surgery; and one or more of the following:

  1. Body mass index ≥ 35 kgm-2
  2. Scoliosis or other spinal deformity
  3. Poorly palpable or impalpable spinous processes

Exclusion Criteria:

* Patient refusal
* Contra-indications to regional anesthesia
* Known allergy to local anesthetics
* Bleeding diathesis
* Inability to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2009-05; Primary Completion 2010-06 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The success rate of dural puncture on the first needle insertion attempt. | within 2 hours prior to surgery

SECONDARY OUTCOMES:
number of needle insertions/re-directions; performance time; Pain score; Patient satisfaction; quality of ultrasound image; Correlation between palpation and ultrasound; Correlation between ultrasound and measured depth to i.t. space | within 2 hours prior to surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ki Jinn Chin, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada